CLINICAL TRIAL: NCT02165735
Title: Addressing HIV Tx Disparities Through Patient Empowerment
Brief Title: Get Ready And Empowered About Treatment
Acronym: GREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Kevin Fiscella, MD, MPH, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AD-1306-03104
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient activation training (Experimental): Patient activation training involves six, 90-minute, group (8-12 person) training sessions facilitated by trained peers and training staff and one (20-30 minute) pre-visit coaching session conducted by staff. The hands on group training includes: 1) HIV education; 2) use of a handheld smart device; 3) use of an HIV electronic personal health record app that runs on the smart device; 4) identification of patients' visit need priorities and skills for communicating with their HIV provider. The pre-visit coaching includes identification patient concerns and patient behavioral rehearsal for asking about these concerns.
  Interventions: Behavioral: patient activation training
- Usual Care (Experimental): Usual care for HIV
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: patient activation training — Patient activation training involves six, 90-minute, group (8-12 person) training sessions facilitated by trained peers and training staff and one (20-30 minute) pre-visit coaching session conducted by staff. The hands on group training includes: 1) HIV education; 2) use of a handheld smart device; 3) use of an HIV electronic personal health record app that runs on the smart device; 4) identification of patients' visit need priorities and skills for communicating with their HIV provider. The pre-visit coaching includes identification of patient concerns and patient behavioral rehearsal for asking about these concerns.
  Arms: patient activation training
Other: Usual care — Usual HIV care
  Arms: Usual Care

SUMMARY:
The purpose of this study is to rigorously assess a program designed to empower patient living with HIV, to improve their health care and health, and to reduce disparities.

DETAILED DESCRIPTION:
Our project has four major aims:

1. Assess improvement in patient empowerment
2. Assess improvement in patients' receipt of evidence-based care
3. Assess improvement in patients' health
4. Assess reduction in disparities in empowerment

ELIGIBILITY:
Inclusion Criteria:

* age18 years or older,
* confirmed HIV diagnosis
* receipt of care within a participating site.

Exclusion Criteria:

* inability to provide informed consent
* limited English proficiency (Trainings and Personal Health Record are currently only available in English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Fiscella, MD MPH, Principal Investigator — University of Rochester; Jonathan Tobin, PhD, Principal Investigator — Clinical Directors Network CDN
Locations (2):
- United States (2):
  - Clinical Directors Network, New York, New York
  - University of Rochester, Rochester, New York

REFERENCES:
- [Derived] Carroll JK, Tobin JN, Luque A, Farah S, Sanders M, Cassells A, Fine SM, Cross W, Boyd M, Holder T, Thomas M, Overa CC, Fiscella K. "Get Ready and Empowered About Treatment" (GREAT) Study: a Pragmatic Randomized Controlled Trial of Activation in Persons Living with HIV. J Gen Intern Med. 2019 Sep;34(9):1782-1789. doi: 10.1007/s11606-019-05102-7. Epub 2019 Jun 25. PMID 31240605
- [Derived] Fiscella K, Boyd M, Brown J, Carroll J, Cassells A, Corales R, Cross W, El'Daher N, Farah S, Fine S, Fowler R, Hann A, Luque A, Rodriquez J, Sanders M, Tobin J. Activation of persons living with HIV for treatment, the great study. BMC Public Health. 2015 Oct 16;15:1056. doi: 10.1186/s12889-015-2382-1. PMID 26474979

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Empowerment: Participants will take part in six 90-minute sessions focused on development of basic information technology competency within a context that supports patient autonomy, competence and human relationships.
  Patient Empowerment and Autonomy Training: Participants will be given supports to address patient autonomy, competence and development of provider-patient relationships.
  Patient Empowerment and Autonomy Training
- Standard Care: Participants will be followed through usual source of care, without receiving the empowerment training.
Period: Overall Study
Arm/Group | Patient Empowerment | Standard Care
Started | 180 | 180
Completed | 164 | 166
Not Completed | 16 | 14
Not completed — Lost to Follow-up | 12 | 10
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Participant indicated lack of time | 1 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: One patient that was randomized to Standard Care was subsequently found to be ineligible for the study. This resulted in 179 participants in the Standard Care arm, rather than 180.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Empowerment | Standard Care | Total
Number analyzed (Participants) | 180 | 179 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.71 (10.71) | 51.24 (11.31) | 51.48 (11)
Sex/Gender, Customized [Number; unit: participants]
  Male | 112 | 101 | 213
  Female | 68 | 75 | 143
  Transgender | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 47 | 83
  Not Hispanic or Latino | 144 | 132 | 276
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 98 | 89 | 187
  White | 43 | 37 | 80
  More than one race | 18 | 12 | 30
  Unknown or Not Reported | 20 | 41 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Activation Measure (PAM)
Description: Our primary outcome measure is patient empowerment based on changes in the Patient Activation Measure or PAM. The Patient Activation Measure (PAM) is a 13-item measure that assesses patient knowledge, skill, and confidence for self-management. People who score high on the PAM normally understand the importance of taking an active role in managing their health and have the skills and confidence to do so.The scores for the 13-item measure range in value from 0-100, with higher scores indicating greater activation.
  LEVEL 1 (0-47): May not yet believe that the patient role is important LEVEL 2 (47.1 - 55.1): Lacks confidence and knowledge to take action LEVEL 3 (55.2 - 67.0): Beginning to take action LEVEL 4 (67.1 - 100): Adapting new behaviors, but may have difficulty maintaining over time
Time Frame: Baseline and 1 year
Population: Multiple imputation was used to account for those with missing or incomplete data
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Patient Empowerment: Participants will take part in six 90-minute sessions focused on development of basic information technology competency within a context that supports patient autonomy, competence and human relationships.
  Patient Empowerment and Autonomy Training: Participants will be given supports to address patient autonomy, competence and development of provider-patient relationships.
Arm/Group | Patient Empowerment | Standard Care
Number analyzed (Participants) | 180 | 179
score on a scale | 73.35 (1.13) | 70.53 (1.14)

2. Secondary Outcome: Change in eHealth Literacy Scale (eHEALS)
Description: Our first secondary outcome measure is eHealth literacy based on changes in the eHealth Literacy Scale or eHEALS. The eHealth Literacy Scale (eHEALS) is an 8-item measure that assesses patient comfort, knowledge, and skills at finding health information on the internet and evaluating whether or not it is reliable. People who score high on the eHEALS normally are very comfortable finding reliable information on the internet. The scores for the 8-item measure range in value from 8-40, with higher scores indicating greater perceived skills at using online health information to help solve health problems.
Time Frame: Baseline and 1 year
Population: Multiple imputation was used to account for those with missing or incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Empowerment | Standard Care
Number analyzed (Participants) | 180 | 179
score on a scale | 29.81 (1.45) | 27.67 (1.42)

3. Secondary Outcome: Change in Decisional Self-Efficacy Scale (DSES)
Description: Our next secondary outcome measure is decision making based on changes in the Decisional Self-Efficacy Scale or DSES. The Decisional Self-Efficacy Scale (DSES) is an 11-item measure that assesses patient confidence in their ability to make health care decisions. People who score high on the DSES normally have an easier time making health care decisions. The scores for the 11-item measure range in value from 0-100, with higher scores indicating greater confidence in making an informed choice.
Time Frame: Baseline and 1 year
Population: Multiple imputation was used to account for those with missing or incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Empowerment | Standard Care
Number analyzed (Participants) | 180 | 179
score on a scale | 91.89 (0.86) | 90.81 (0.87)

4. Secondary Outcome: Change in Perceived Involvement in Care Scale (PICS)
Description: Our third secondary outcome measure is involvement in care based on changes in the Perceived Involvement in Care Scale or PICS. The Perceived Involvement in Care Scale (PICS) is an 8-item measure that assesses patient perceived proficiency in communicating concerning their health care with the doctor. People who score high on the PICS normally are satisfied with how well they feel they communicate with the doctor about their care. The scores for the 8-item measure range in value from 8-40, with higher scores indicating greater perceived involvement in their care.
Time Frame: Baseline and 1 year
Population: Multiple imputation was used to account for those with missing or incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Empowerment | Standard Care
Number analyzed (Participants) | 180 | 179
score on a scale | 33.74 (0.94) | 32.47 (0.90)

5. Secondary Outcome: Change in Instrument on Doctor Patient Communication Skills (IDPCS)
Description: Our fourth secondary outcome measure is clinician patient centeredness based on changes in the Instrument on Doctor Patient Communication Skills or IDPCS. The Instrument on Doctor Patient Communication Skills (IDPCS) is a 19-item measure that assesses patient perception of the doctor's communication proficiency with them. People who score high on the IDPCS normally are satisfied with the way the doctor speak with them about their care. The scores for the 19-item measure range in value from 19-95, with higher scores indicating greater quality communication by the doctor.
Time Frame: Baseline and 1 year
Population: Multiple imputation was used to account for those with missing or incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Empowerment | Standard Care
Number analyzed (Participants) | 180 | 179
score on a scale | 85.06 (1.24) | 83.49 (1.25)

6. Secondary Outcome: Change in HIV Adherence Self-Efficacy Scale (ASES)
Description: Our fifth secondary outcome measure is HIV adherence self-efficacy based on changes in the HIV Adherence Self-Efficacy Scale or ASES. The HIV Adherence Self-Efficacy Scale (ASES) is a 15-item measure that assesses patient self-efficacy for adherence to HIV treatment plan including but not limited to taking HIV medications. People who score high on the ASES normally are very confident of sticking to their HIV treatment plan even when it is hard. The scores for the 15-item measure range in value from 0-150, with higher scores indicating greater adherence self-efficacy.
Time Frame: Baseline and 1 year
Population: Multiple imputation was used to account for those with missing or incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Empowerment | Standard Care
Number analyzed (Participants) | 180 | 179
score on a scale | 102.80 (1.08) | 103.13 (1.07)

7. Secondary Outcome: Change in Self-Reported Adherence
Description: Our sixth secondary outcome measure is adherence to combination antiretroviral treatment (cART) based on changes on survey of recommended items for assessing self-reported antiretroviral adherence. Our survey included two recommended assessment items with the focus on one-item measure that assesses patient self-reported adherence to taking HIV medications. People who score high on the self-reported adherence cART normally are very confident of being more adherent to taking their HIV medications. The score for the one-item measure range in value from 0-100 percent, with higher scores indicating greater adherence to cART.
Time Frame: Baseline and 1 year
Population: Multiple imputation was used to account for those with missing or incomplete data.
Measure: Mean (Standard Deviation); unit: percentage of cART adherence in past mth
Arm/Group | Patient Empowerment | Standard Care
Number analyzed (Participants) | 180 | 179
percentage of cART adherence in past mth | 89.33 (1.09) | 89.90 (1.09)

8. Secondary Outcome: Change in Undetectable Viral Load
Description: Our seventh secondary outcome measure is undetectable viral load based on changes to participants' HIV viral load. The HIV viral load measurements were abstracted from the participants' personal health record (PHR). In our study, people who had a HIV viral load of <50 were considered to have undetectable viral load.
Time Frame: Baseline and 1 year
Population: Multiple imputation was used to account for those with missing or incomplete data.
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Patient Empowerment | Standard Care
Number analyzed (Participants) | 180 | 179
percentage of participants | 87 (3.1) | 86 (3.1)

9. Secondary Outcome: Change in Evidence-based Preventative Care
Description: Our eighth secondary outcome measure is prevention-seeking behavior based on chart abstracted information based on our preventive care index. We created a preventive care index for each participant by assigning one point of each intervention they received post-randomization divided by the total number of interventions for which they were eligible. The index included eleven preventive care measures: Human Papillomavirus, Influenza, Tetanus, Hepatitis A, B, C testing, Hepatitis A & B vaccinations, cervical cancer screening (PAP), mammography and any colon cancer screening. People who score high on the evidence-based preventative care normally are more able to prevent illnesses or diseases. The score for the measure range in value from 0-1, with higher scores indicating greater ability to stay healthy.
Time Frame: Baseline and 1 year
Population: Multiple imputation was used to account for those with missing or incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Empowerment | Standard Care
Number analyzed (Participants) | 180 | 179
score on a scale | 0.35 (0.01) | 0.35 (0.02)

10. Secondary Outcome: Change in Short Form Health Survey: [Mental Health] (SF12)
Description: Our ninth secondary outcome measure is mental well-being and quality of life based on changes on the Short Form Health Survey or SF12. The Short Form Health Survey (SF12) is a 12-item measure with 6 items that assesses patient mental well-being/quality of life and 6 items that assesses patient physical well-being/quality of life. People who score high on the SF-12 are normally in good mental and physical health. The scores for the 12-item measure includes two scales whose range in value from 0-100, with higher scores indicating a better health state.
Time Frame: Baseline and 1 year
Population: Multiple imputation was used to account for those with missing or incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Empowerment | Standard Care
Number analyzed (Participants) | 180 | 179
score on a scale | 46.38 (0.73) | 46.99 (0.73)

11. Secondary Outcome: Change in Short Form Health Survey: [Physical Health] (SF12)
Description: Our final secondary outcome measure is physical well-being and quality of life based on changes on the Short Form Health Survey or SF12. The Short Form Health Survey (SF12) is a 12-item measure with 6 items that assesses patient mental well-being/quality of life and 6 items that assesses patient physical well-being/quality of life. People who score high on the SF-12 are normally in good mental and physical health. The scores for the 12-item measure includes two scales whose range in value from 0-100, with higher scores indicating a better health state.
Time Frame: Baseline and 1 year
Population: Multiple imputation was used to account for those with missing or incomplete data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Empowerment | Standard Care
Number analyzed (Participants) | 180 | 179
score on a scale | 44.83 (0.71) | 45.13 (0.72)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Patient Empowerment | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/180
Serious Adverse Events (participants affected / at risk) | 0/180 | 0/180
Other Adverse Events (participants affected / at risk) | 0/180 | 0/180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No